CLINICAL TRIAL: NCT00581165
Title: Evaluating Safety in Patients With Moderate to Severe Psoriasis Treated With Etanercept
Brief Title: Study Evaluating Safety of Etanercept in Treatment of Patients With Moderate to Severe Psoriasiswith Etanercept
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinial Trials Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0881A1-101781
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Etanercept — recommended dose of enbrel is 25mg administered twice weekly.

SUMMARY:
Evaluate (i) safety of etanercept in patients with moderate to severe psoriasis in Spain; (ii) the incidence of adverse events reported in these patients, and (iii) the role that age and concomitant therapy might play in the development of adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed by patients prior to study entry
2. 18 years of age or older at screening visit
3. Patients with moderate to severe psoriasis
4. Patients who have failed conventional systemic treatment
5. Patients who have a contraindication to conventional systemic therapy
6. Patients who are intolerant to conventional systemic therapy
7. A negative serum pregnancy test at screening in women of childbearing potential
8. Able to self-inject study drug or have a designee who can do so
9. In the opinion of the investigator, the patient will be able to comply with the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2006-02; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Dermatology Quality of Life Index, Psoriasis Quality of Life Index and Physician Global assessment | 18 months

SECONDARY OUTCOMES:
Reduction and/or withdrawal of systemic therapies, Proportion of patients with plaque psoriasis achieving PASI 50, 75 and 90 at each evaluation and BSA at each evaluation | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer